CLINICAL TRIAL: NCT02682732
Title: Molecular Imaging to Capture Disease Heterogeneity in Acute Myeloid Leukemia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hamilton Health Sciences Corporation (Other)
Responsible Party: Principal Investigator, Mohammed Almakadi, MBBS, FRCP(C), Hamilton Health Sciences Corporation
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: NIF-15378
Record Dates: First submitted 2016-02-03; First posted 2016-02-15 (Estimated); Last update posted 2018-02-22 (Actual); Status verified 2018-02

CONDITIONS: Leukemia, Myeloid, Acute
Keywords: Acute Myeloid Leukemia; PET/CT Scan
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- FDG-PET/CT (Experimental): (Fluorodeoxyglucose positron-emission tomography) FDG-PET/CT guided bone marrow sampling will be performed at diagnosis and at the end of induction chemotherapy (like cytarabine and daunorubicin). Then, patients will be followed to assess their response, and imaging-guided bone marrow sampling will be repeated in the likely event of disease relapse.
  Interventions: Procedure: FDG-PET/CT guided bone marrow sampling

INTERVENTIONS:
Procedure: FDG-PET/CT guided bone marrow sampling — (Fluorodeoxyglucose positron-emission tomography) FDG-PET/CT guided bone marrow sampling will be used to obtain two different samples from avid and dim bone marrow areas.

SUMMARY:
The current understanding of acute myeloid leukemia (AML) is that one site of bone marrow (BM) sampling serves as a window that represents all AML cells distributed throughout the BM, an assumption that has yet to be questioned. Simulation in mice led to inconsistent representation of the full BM, which can incorrectly suggest the absence of leukemic cells. Positron-emission tomography (PET) scan can detect areas of high metabolic activity in the body using for instance a radioactive sugar. In one report, its use in human AML has provided proof-of-principle evidence of unequal distribution of AML cells in BM. Accordingly, the alternative hypothesis is to test if PET scan can demonstrate if BM geography can alter AML cells spread and home them as distinct areas rather than uniform spread as if they are distributed in liquid state.

ELIGIBILITY:
Inclusion Criteria:

* New diagnosis of AML according to the WHO (World Health Organization) criteria

Exclusion Criteria:

* Prior malignancy, unless the patient has been disease-free for at least five years following curative intent therapy, with the following exceptions: patients with treated non-melanoma skin cancer, in situ carcinoma, or cervical intraepithelial neoplasia, regardless of the disease-free duration, if definitive treatment for the condition has been completed; or patients with organ-confined prostate cancer with no evidence of recurrent or progressive disease.
* Acute promyelocytic leukemia (APL).
* ECOG (Eastern Cooperative Oncology Group) performance status of 3 or more
* Inadequate renal function (i.e., estimated GFR (glomerular filtration rate) < 60 mL/min/1.73m2).
* Inadequate hepatic function (i.e., serum bilirubin > 1.5×ULN; AST (aspartate aminotransferase), ALT (alanine aminotransferase) and ALP (alkaline phosphatase) > 2.5×ULN)
* Presence of uncontrolled systemic fungal, bacterial, viral or other infections (defined as exhibiting ongoing signs/symptoms related to the infection and without improvement, despite appropriate antibiotics or other treatment).
* Having any other severe concurrent disease or serious organ dysfunction that may place the patient at undue risk to receive induction therapy.
* Pregnancy or lactating female.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2016-04; Primary Completion 2019-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Number of patients with heterogeneous (positron-emission tomography) PET/CT activity before induction chemotherapy | Up to 3 years

SECONDARY OUTCOMES:
Number of patients with residual (positron-emission tomography) PET/CT activity following induction chemotherapy | Up to 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Mickie Bhatia, PhD, Study Director — McMaster University
Locations (1):
- Juravinski Hospital and Cancer Center, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
The data will be shared after the study is completed

REFERENCES:
- See also: Acute Myeloid Leukemia — https://www.nlm.nih.gov/medlineplus/acutemyeloidleukemia.html
- See also: PET Scan — https://www.nlm.nih.gov/medlineplus/ency/article/003827.htm